CLINICAL TRIAL: NCT07268833
Title: Translating Single-cell Vulnerability Into Novel ALS Biomarkers and Therapeutic Targets: Towards a Liquid Nerve Biopsy
Acronym: TUNEABLE
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: Azienda Ospedaliero Universitaria di Cagliari (Other); IRCCS San Raffaele (Other); Università di Napoli Federico II (Unknown)
Responsible Party: Sponsor
Other Study IDs: PNRR-MCNT2-2023-12377651
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS); Peripheral Neuropathies
Keywords: ALS; Peripheral Neuropathies; Motor Neuron Disease; Biomarkers; Neurodegeneration; Nerve Biopsy; skin biopsy; Spatial Transcriptomics
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Peripheral Nervous System Diseases; Motor Neuron Disease; Nerve Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1: ALS patients
- 2: Neuropathy patients
- 3: presymptomatic patients
- 4: healthy controls
- 5: Other neurodegenerative diseases

SUMMARY:
The progress of ALS research and clinical practice is hampered by lack of effective biomarkers to monitor disease onset and progression. In response to this urgent need, we will integrate single-cell system biology approaches, histopathological and clinical data from precious human nerve biopsies collected from living ALS patients during the diagnostic workup and findings from innovative preclinical mouse models to unmask cell-specific molecular alterations that arise in the PNS tissue during the course of ALS pathology. This information will be used to select protein biomarkers of dysfunctional states associated with pre-manifest or early symptomatic stages of the disease, which will be further screened and validated in patient biofluids. Altogether, this project will lead to the discovery of novel, reliable and specific ALS biomarkers while providing insights into ALS mechanisms by leveraging an original "PNS perspective" on disease pathogenesis.

DETAILED DESCRIPTION:
The absence of specific biomarkers poses a significant impediment to the advancement of new treatments for amyotrophic lateral sclerosis (ALS), a severe and rapidly fatal neurodegenerative disease with no cure to date, defined by degeneration of motor neurons. Early pathological events, such as the selective damage of motor axons and the loss of neuromuscular connections, precede complete neurodegeneration and the manifestation of clinical symptoms. Therefore, we argue that understanding disease-related changes occurring in peripheral nerves is crucial for defining the underlying pathogenetic mechanisms. Preliminary data from our research team suggest that phosphorylated TDP-43, the pathological hallmark of ALS, forms aggregates in motor axons and Schwann cells of living ALS patients before the onset of axonal degeneration. However, peripheral nerves constitute complex multicellular tissues, and the specific contributions of individual cellular components to ALS pathology remain poorly understood. The overarching concept of this proposal is that distinct cell types within the nerve tissue (e.g., Schwann cells, endothelial cells, fibroblasts, macrophages) function as exquisite early detectors of motor neuron damage and initiate secondary responses that amplify neuropathology. These studies will steer the analysis of minimally invasive skin biopsies to uncover deregulated PNS signatures in ALS patients. Finally, candidate molecular targets reflecting cell-type-specific deregulation in the diseased nerve microenvironment will be screened in the biofluids of ALS patients and at-risk individuals from genetic ALS families, enabling the discovery of novel diagnostic and prognostic biomarkers. The integrative approach proposed in this study will elucidate the pathogenic mechanisms of ALS and establish a roadmap towards identifying potential therapeutic targets.

ELIGIBILITY:
Inclusion Criteria for als patients:

* Age equal or over 18 years old
* ALS patients, diagnosed accordingly to the revised El Escorial Criteria
* Disease duration <24 months from symptom onset.

Exclusion Criteria for als patients:

* FVC <60%;
* nutritional or respiratory failure;
* significant hepatic or chronic renal failure or any interveninginfective or metabolic conditions potentially influencing CBs levels.

Inclusion criteria for ALS pre-symptomatic patients

* Age equal or over 18 years old
* Patients with genetic defined susceptibility to ALS and one or more strict relative affected from ALS Exclusion criteria for ALS pre-symptomatic patients
* significant hepatic or chronic renal failure or any interveninginfective or metabolic conditions potentially influencing CBs levels.

Inclusion criteria for controls

* Age equal or over 18 years old
* Subjects without a diagnosis of neurodegenerative disease or neuromuscular disorder.

Exclusion criteria for controls

• significant hepatic or chronic renal failure or any interveninginfective or metabolic conditions potentially influencing CBs levels.

Inclusion criteria for non ALS neurodegenerative patients

* Age equal or over 18 years old
* For AD: Diagnosis according to 2018 NIA-AA Framework for Alzheimer's Disease
* For FTD: Diagnosis according to 2011 International Behavioural Variant FTD Criteria Consortium
* For PD: Diagnosis according to 2015 Movement Disorder Society criteria
* For DLB: Diagnosis according to 2017 Fourth Consensus Report of the DLB Consortium Exclusion criteria for non ALS neurodegenerative patients
* significant hepatic or chronic renal failure or any interveninginfective or metabolic conditions potentially influencing CBs levels.

Inclusion criteria for neuromuscular disease patients

* Age equal or over 18 years old
* Presence of axonal or demyelinating neuropathy Exclusion criteria for neuromuscular patients
* significant hepatic or chronic renal failure or any interveninginfective or metabolic conditions potentially influencing CBs levels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Number of patients projected for:
  * the entire study: 400 patients
  * each treatment group: ALS 150, HC 40, non-ALS neurodegenerative 60, non-ALS neuromuscular diseases 50, Indipendent cohort of ALS Sardinian patients 100.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic ALS biomarkers | 20 months
  Throughout the study, we will validate, starting from transcriptomics data, novel diagnostic biomarker for an early diagnosis of ALS

SECONDARY OUTCOMES:
Prognostic biomarkers | 24 months
  explore novel prognostic biomarkers, able to reliably predict the time-course of ALS
Therapeutic targets | 24 months
  identify molecular targets related to axonal degeneration for potential therapeutic intervention

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Azienda Ospedaliero Universitaria di Cagliari, Monserrato, California
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - IRCCS Ospedale San Raffaele SRL, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli

REFERENCES:
- [Background] Rocha MC, Pousinha PA, Correia AM, Sebastiao AM, Ribeiro JA. Early changes of neuromuscular transmission in the SOD1(G93A) mice model of ALS start long before motor symptoms onset. PLoS One. 2013 Sep 5;8(9):e73846. doi: 10.1371/journal.pone.0073846. eCollection 2013. PMID 24040091
- [Background] Riva N, Iannaccone S, Corbo M, Casellato C, Sferrazza B, Lazzerini A, Scarlato M, Cerri F, Previtali SC, Nobile-Orazio E, Comi G, Quattrini A. Motor nerve biopsy: clinical usefulness and histopathological criteria. Ann Neurol. 2011 Jan;69(1):197-201. doi: 10.1002/ana.22110. Epub 2010 Nov 12. PMID 21280090
- [Background] Riva N, Gentile F, Cerri F, Gallia F, Podini P, Dina G, Falzone YM, Fazio R, Lunetta C, Calvo A, Logroscino G, Lauria G, Corbo M, Iannaccone S, Chio A, Lazzerini A, Nobile-Orazio E, Filippi M, Quattrini A. Phosphorylated TDP-43 aggregates in peripheral motor nerves of patients with amyotrophic lateral sclerosis. Brain. 2022 Mar 29;145(1):276-284. doi: 10.1093/brain/awab285. PMID 35076694
- [Background] Riva N, Clarelli F, Domi T, Cerri F, Gallia F, Trimarco A, Brambilla P, Lunetta C, Lazzerini A, Lauria G, Taveggia C, Iannaccone S, Nobile-Orazio E, Comi G, D'Antonio M, Martinelli-Boneschi F, Quattrini A. Unraveling gene expression profiles in peripheral motor nerve from amyotrophic lateral sclerosis patients: insights into pathogenesis. Sci Rep. 2016 Dec 16;6:39297. doi: 10.1038/srep39297. PMID 27982123
- [Background] Nolano M, Provitera V, Manganelli F, Iodice R, Caporaso G, Stancanelli A, Marinou K, Lanzillo B, Santoro L, Mora G. Non-motor involvement in amyotrophic lateral sclerosis: new insight from nerve and vessel analysis in skin biopsy. Neuropathol Appl Neurobiol. 2017 Feb;43(2):119-132. doi: 10.1111/nan.12332. Epub 2016 Jul 7. PMID 27288647
- [Background] Gentile F, Scarlino S, Falzone YM, Lunetta C, Tremolizzo L, Quattrini A, Riva N. The Peripheral Nervous System in Amyotrophic Lateral Sclerosis: Opportunities for Translational Research. Front Neurosci. 2019 Jun 25;13:601. doi: 10.3389/fnins.2019.00601. eCollection 2019. PMID 31293369
- [Background] Fischer LR, Culver DG, Tennant P, Davis AA, Wang M, Castellano-Sanchez A, Khan J, Polak MA, Glass JD. Amyotrophic lateral sclerosis is a distal axonopathy: evidence in mice and man. Exp Neurol. 2004 Feb;185(2):232-40. doi: 10.1016/j.expneurol.2003.10.004. PMID 14736504
- [Background] Casiraghi V, Milone I, Brusati A, Peverelli S, Doretti A, Poletti B, Maderna L, Morelli C, Ticozzi N, Silani V, Verde F, Ratti A. Quantification of serum TDP-43 and neurofilament light chain in patients with amyotrophic lateral sclerosis stratified by UNC13A genotype. J Neurol Sci. 2024 Nov 15;466:123210. doi: 10.1016/j.jns.2024.123210. Epub 2024 Sep 2. PMID 39241471
- [Background] Brodovitch A, Boucraut J, Delmont E, Parlanti A, Grapperon AM, Attarian S, Verschueren A. Combination of serum and CSF neurofilament-light and neuroinflammatory biomarkers to evaluate ALS. Sci Rep. 2021 Jan 12;11(1):703. doi: 10.1038/s41598-020-80370-6. PMID 33436881
- [Background] Bhat GP, Maurizio A, Motta A, Podini P, Diprima S, Malpighi C, Brambilla I, Martins L, Badaloni A, Boselli D, Bianchi F, Pellegatta M, Genua M, Ostuni R, Del Carro U, Taveggia C, de Pretis S, Quattrini A, Bonanomi D. Structured wound angiogenesis instructs mesenchymal barrier compartments in the regenerating nerve. Neuron. 2024 Jan 17;112(2):209-229.e11. doi: 10.1016/j.neuron.2023.10.025. Epub 2023 Nov 15. PMID 37972594
- [Background] Barrientos SA, Martinez NW, Yoo S, Jara JS, Zamorano S, Hetz C, Twiss JL, Alvarez J, Court FA. Axonal degeneration is mediated by the mitochondrial permeability transition pore. J Neurosci. 2011 Jan 19;31(3):966-78. doi: 10.1523/JNEUROSCI.4065-10.2011. PMID 21248121